CLINICAL TRIAL: NCT04190056
Title: Epigenetic Priming for Immune Therapy in ER-Positive Breast Cancer in Biomarker Select Population
Brief Title: Pembrolizumab and Tamoxifen With or Without Vorinostat for the Treatment of Estrogen Receptor Positive Breast Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Change in practice patterns
Sponsor: University of California, San Francisco (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 197520; NCI-2019-07572 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2019-12-04; First posted 2019-12-09 (Actual); Results first posted 2023-08-31 (Actual); Last update posted 2023-08-31 (Actual); Status verified 2023-08

CONDITIONS: Anatomic Stage IV Breast Cancer AJCC v8; Prognostic Stage IV Breast Cancer AJCC v8
MeSH Terms: interventions — pembrolizumab; Tamoxifen; Vorinostat

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm A (pembrolizumab, vorinostat, tamoxifen) (Experimental): Patients receive pembrolizumab IV over 30 minutes on day 1, vorinostat PO QD for 4 days weekly, and tamoxifen PO QD on days 1-21. Cycles repeat every 21 days in the absence of disease progression of unacceptable toxicity.
  Interventions: Biological: Pembrolizumab; Drug: Tamoxifen; Drug: Vorinostat
- Arm B (pembrolizumab, tamoxifen) (Experimental): Patients receive pembrolizumab IV over 30 minutes on day 1 and tamoxifen PO QD on days 1-21. Cycles repeat every 21 days in the absence of disease progression of unacceptable toxicity.
  Interventions: Biological: Pembrolizumab; Drug: Tamoxifen

INTERVENTIONS:
Biological: Pembrolizumab — Given IV
  Other Names: Keytruda; Lambrolizumab; MK-3475; SCH 900475
Drug: Tamoxifen — Given PO
Drug: Vorinostat — Given PO
  Other Names: L-001079038; MSK-390; SAHA; Suberanilohydroxamic Acid; Suberoylanilide Hydroxamic Acid; Zolinza
  Arms: Arm A (pembrolizumab, vorinostat, tamoxifen)

SUMMARY:
This phase II trial studies how well pembrolizumab and tamoxifen with or without vorinostat work for the treatment of estrogen receptor positive breast cancer. Immunotherapy with monoclonal antibodies, such as pembrolizumab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread. Estrogen can cause the growth of breast cancer cells. Hormone therapy with tamoxifen may may fight breast cancer by blocking the use of estrogen by the tumor cells. Vorinostat may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. This trial is being done to find a drug combination to better control estrogen receptor positive breast cancer and reduce the number of pills taken.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To define the role of epigenetic immune priming in a biomarker enriched estrogen receptor (ER)+ breast cancer population on the basis of overall response rate.

SECONDARY OBJECTIVES:

I. To assess duration of response (DOR) 24-week landmark progression-free survival (PFS:24).

II. Median PFS and overall survival (OS). III. Tumor responses will also be calculated by Immune Related Response-Criteria (irRC).

EXPLORATORY OBJECTIVES:

I. Evaluation of biomarker target threshold on response rate (retrospective cut off of 20% versus [vs] 10%).

II. To assess the ratio of effector T cells: regulatory T cells in blood and tumor biopsies pre- and post-therapy.

III. To evaluate inflammatory T cell signature changes in blood and tumor biopsies pre- and post-therapy.

IV. To evaluate changes in number of myeloid-derived suppressor cells (MDSCs) in peripheral blood and tumor biopsies pre- and posttherapy.

V. To evaluate changes in histone acetylation in peripheral blood cells and tumor biopsies pre- and post-therapy.

VI. Initial comparison to vorinostat-induced PD-1 in lymphocytes, PD-L1 modulation.

VII. Nanostring and 10 x sequencing and single cell immune phenotyping (on stored tissue for successful arms only).

VIII. Impact of histone deacetylase (HDAC) inhibition of response to pembrolizumab vs. pembrolizumab in biomarker enriched population.

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM A: Patients receive pembrolizumab intravenously (IV) over 30 minutes on day 1, vorinostat orally (PO) once daily (QD) for 4 days weekly, and tamoxifen PO QD on days 1-21. Cycles repeat every 21 days in the absence of disease progression of unacceptable toxicity.

ARM B: Patients receive pembrolizumab IV over 30 minutes on day 1 and tamoxifen PO QD on days 1-21. Cycles repeat every 21 days in the absence of disease progression of unacceptable toxicity.

After completion of study treatment, patients are followed up for 30 days and then every 12 weeks thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Pre and postmenopausal women or men with stage IV ER+ breast cancer histological or cytological confirmation
* > 10% expression of PD-1/Cytotoxic T-lymphocyte-associated protein 4 (CTLA-4) dual staining in Cluster of differentiation 8 (CD8) cells in tumor or blood or >5% expression of PD-1/CTLA-4 dual staining in CD4 in blood (only).
* Eastern Cooperative Oncology Group (ECOG) performance status of =< 1
* Understand and voluntarily sign an informed consent prior to any study-related assessments or procedures are conducted and are able to adhere to the study visit schedule and other protocol requirements
* Consent to paired tumor biopsy
* Measurable tumor by Response Evaluation Criteria in Solid Tumors (RECIST) criteria
* Per Good Clinical Practice, any toxicity related to prior therapies that, in the opinion of the investigator, would potentially be worsened with anti-PD1 therapy should be resolved to less than grade 1
* Absolute neutrophil count (ANC) >= 1.5 X 10^9/L
* Hemoglobin (Hgb) >= 9 g/dL (may transfuse if clinically indicated)
* Platelets (plt) >= 100 x 10^9/L
* Potassium within normal range, or correctable with supplements
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) =< 2.5 x upper limit normal (ULN) or =< 5.0 x ULN if liver tumor is present
* Serum total bilirubin =< 1.5 x ULN
* Serum creatinine =< 1.5 x ULN, or 24-hr clearance >= 60 ml/min
* Females of childbearing potential (defined as sexually mature women who):

  * Has not undergone a hysterectomy (the surgical removal of the uterus) or bilateral oophorectomy (the surgical removal of both ovaries) or,
  * Has not been naturally postmenopausal for at least 24 consecutive months (i.e., has had menses at any time during the preceding 24 consecutive months) must have

    * Negative serum pregnancy test within 14 days before starting study treatment in females of childbearing potential (FCBP) and willingness to adhere to acceptable forms or birth control (a physician-approved contraceptive method (oral, injectable, or implantable hormonal contraceptive; tubal ligation; intra-uterine device; barrier contraceptive with spermicide; or vasectomized partner)
* All female and male participants must agree to use approved contraception during the treatment period and for at least 18 weeks after the last dose of study treatment and refrain from donating sperm during this period

Exclusion Criteria:

* Prior treatment with pembrolizumab or other PD-(L)1
* Any significant medical condition, laboratory abnormalities, which places the subject at unacceptable risk if he/she were to participate in the study
* Has a history of (non-infectious) pneumonitis/interstitial lung disease that required steroids or current pneumonitis/ interstitial lung disease
* Has known active hepatitis B (e.g., hepatitis B surface antigen (HBsAg) reactive) or hepatitis C (e.g., hepatitis C virus (HCV) ribonucleic acid (RNA) [qualitative] is detected)
* Has a history of hepatitis B virus (HBV)
* Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the study, interfere with the subject's participation for the full duration of the study, or is not in the best interest of the subject to participate, in the opinion of the treating investigator
* Symptomatic central nervous system metastases. Subjects with brain metastases that have been previously treated and are stable for 6 weeks are allowed
* Persistent diarrhea or malabsorption >= National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) grade 2, despite medical management
* Unstable angina, significant cardiac arrhythmia, or New York Heart Association (NYHA) class 3 or 4 congestive heart failure
* Prior systemic cancer-directed treatments or investigational modalities =< 5 half-lives or 4 weeks, whichever is shorter, prior to starting study drug or who have not recovered from side effects of such therapy (except alopecia)
* Active autoimmune disease except for vitiligo or hypothyroidism
* Active and ongoing steroid use, except for non-systemically absorbed treatments (such as inhaled or topical steroid therapy for asthma, chronic obstructive pulmonary disease (COPD), allergic rhinitis)
* Major surgery =< 2 weeks prior to starting a study drug or who have not recovered from side effects of such therapy
* Pregnant or breastfeeding
* Known human immunodeficiency virus (HIV) infection
* Known history of tuberculosis
* Known allergic reaction or intolerability to tamoxifen
* Patients with prior history of deep vein thrombosis (DVT)s must be on therapeutic or preventive anticoagulation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2021-03-11 (Actual); Primary Completion 2023-06-15 (Actual); Study Completion 2023-06-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pamela Munster, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm A (Pembrolizumab, Vorinostat, Tamoxifen): Patients receive pembrolizumab IV over 30 minutes on day 1, vorinostat given orally (PO) every day (QD) for 4 days weekly, and tamoxifen PO QD on days 1-21. Cycles repeat every 21 days in the absence of disease progression of unacceptable toxicity.
Period: Overall Study
Arm/Group | Arm A (Pembrolizumab, Vorinostat, Tamoxifen) | Arm B (Pembrolizumab, Tamoxifen)
Started | 0 | 1
Completed | 0 | 1
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: The study closed early due to a change in practice patterns, and no participants were enrolled on arm A
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A (Pembrolizumab, Vorinostat, Tamoxifen) | Arm B (Pembrolizumab, Tamoxifen) | Total
Number analyzed (Participants) | 0 | 1 | 1
Age, Customized [Count of Participants; unit: Participants] — Year range provided to lessen the probability of a HIPAA violation in public reporting of single participant study
  Participants
    50-59 years | 0 | 1 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 1
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 0 | 1 | 1
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 1 | 1
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States |  | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate (ORR)
Description: ORR is defined as the proportion of participants randomized to that arm whose status is stable disease (SD) or better (complete response (CR), partial response (PR)). Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions: CR=Disappearance of all target lesions; PR = >=30% decrease in the sum of the longest diameter of target lesions, and SD=Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for progressive disease,.
Time Frame: Up to 24 weeks
Population: No participants were enrolled in Arm A
Measure: Number; unit: proportion of participants
Arm/Group | Arm A (Pembrolizumab, Vorinostat, Tamoxifen) | Arm B (Pembrolizumab, Tamoxifen)
Number analyzed (Participants) | 0 | 1
proportion of participants |  | 0

2. Secondary Outcome: Percentage of Participants With Tumor Responses
Description: Tumor responses will be classified using the Immune Related Response-Criteria (irRC)) through study completion.
Time Frame: Up to 24 months
Population: No participants were enrolled in Arm A.
Measure: Number; unit: percentage of participants
Arm/Group | Arm A (Pembrolizumab, Vorinostat, Tamoxifen) | Arm B (Pembrolizumab, Tamoxifen)
Number analyzed (Participants) | 0 | 1
percentage of participants |  | 0

3. Secondary Outcome: Duration of Response (DOR)
Description: The duration of overall response is measured from the time measurement criteria are met for CR or PR (whichever is first recorded) until the first date that recurrent or progressive disease is objectively documented (taking as reference for progressive disease the smallest measurements recorded since the treatment started). The duration of overall CR is measured from the time measurement criteria are first met for CR until the first date that recurrent disease is objectively documented. Duration of stable disease is measured from the start of the treatment until the criteria for progression are met, taking as reference the smallest measurements recorded since the treatment started. Will use median DOR (computed by the Kaplan-Meier estimator) to summarize. The respective confidence intervals will be computed as well.
Time Frame: Up to 24 weeks
Population: No participants were enrolled in Arm A
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Arm A (Pembrolizumab, Vorinostat, Tamoxifen) | Arm B (Pembrolizumab, Tamoxifen)
Number analyzed (Participants) | 0 | 1
weeks |  | NA [NA to NA] — Participant did not have objective response so duration of response cannot be calculated

4. Secondary Outcome: Median Progression Free Survival (PFS)
Description: Progression-free survival (PFS) is defined as the duration of time from start of treatment to time of progression or death from any cause on study, whichever occurs first. Will use median PFS (computed by the Kaplan-Meier estimator) to summarize. The respective confidence intervals will be computed as well.
Time Frame: Up to 27 months
Population: No participants were enrolled in Arm A
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm A (Pembrolizumab, Vorinostat, Tamoxifen) | Arm B (Pembrolizumab, Tamoxifen)
Number analyzed (Participants) | 0 | 1
months |  | NA [NA to NA] — Insufficient number of participants with events

5. Secondary Outcome: Median Overall Survival (OS)
Description: Will use median OS (computed by the Kaplan-Meier estimator) to summarize from initiation of study treatment to the time of death from any cause on study. The respective confidence intervals will be computed as well.
Time Frame: Up to 27 months
Population: No participants were enrolled in Arm A
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm A (Pembrolizumab, Vorinostat, Tamoxifen) | Arm B (Pembrolizumab, Tamoxifen)
Number analyzed (Participants) | 0 | 1
months |  | NA [NA to NA] — Insufficient number of participants with events

ADVERSE EVENTS:
Time Frame: Up to 27 months
Description: No participants were enrolled in Arm A.
Arm/Group | Arm A (Pembrolizumab, Vorinostat, Tamoxifen) | Arm B (Pembrolizumab, Tamoxifen)
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/1
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/1
Other Adverse Events (participants affected / at risk) | 0/0 | 0/1

LIMITATIONS AND CAVEATS:
The study closed early due to change in practice patterns

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-09-30): https://cdn.clinicaltrials.gov/large-docs/56/NCT04190056/Prot_SAP_000.pdf
  • Informed Consent Form (2023-01-05): https://cdn.clinicaltrials.gov/large-docs/56/NCT04190056/ICF_001.pdf